CLINICAL TRIAL: NCT00304005
Title: A Phase I/II Study of Cloretazine in Patients With Refractory/Relapsed Chronic Lymphocytic Leukemia or Richter's Syndrome
Brief Title: VNP40101M in Treating Patients With Richter Syndrome or Refractory or Relapsed Chronic Lymphocytic Leukemia or Other Lymphoproliferative Disorders
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vion Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: VION-CLI-041; CDR0000465217 (Registry Identifier: PDQ (Physician Data Query)); MDA-2005-0249
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2008-08

CONDITIONS: Leukemia; Lymphoma
Keywords: refractory chronic lymphocytic leukemia; recurrent adult diffuse large cell lymphoma; recurrent adult Hodgkin lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Hodgkin Disease | interventions — laromustine

INTERVENTIONS:
Drug: laromustine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as VNP40101M, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase I/II trial is studying the side effects and best dose of VNP40101M and to see how well it works in treating patients with Richter syndrome or refractory or relapsed chronic lymphocytic leukemia or other lymphoproliferative disorders.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose (MTD) of VNP40101M in patients with Richter syndrome or refractory or relapsed chronic lymphocytic leukemia or other lymphoproliferative disease. (phase I)
* Determine the toxic effects of this drug in these patients. (phase I)
* Determine the efficacy, as determined by overall response rate, of this drug at the MTD determined in phase I in these patients. (phase II)

OUTLINE: This is a phase I dose-escalation study followed by a phase II study.

* Phase I: Patients receive VNP40101M IV over 30 minutes on day 1. Courses repeat every 3-6 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of VNP40101M until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

* Phase II: Patients receive VNP40101M at the MTD determined in phase I.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following hematologic malignancies:

  * Fludarabine refractory or relapsed chronic lymphocytic leukemia (CLL)

    * CLL in transformation allowed
  * Richter syndrome
  * Other refractory lymphoproliferative diseases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Creatinine ≤ 2.0 mg/dL

  * Renal dysfunction due to organ infiltration by disease allowed
* AST and ALT ≤ 3 times upper limit of normal (ULN) (unless due to organ infiltration by disease)
* Bilirubin ≤ 1.5 times ULN (unless due to Gilbert's syndrome)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection
* No symptomatic coronary artery disease
* No arrhythmia not controlled by medication
* No uncontrolled, symptomatic congestive heart failure
* No myocardial infarction within the past 3 months
* No other uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

* At least 2 weeks since prior cytotoxic therapy except in patients with rapidly progressing disease
* No other concurrent standard or investigational treatment for this cancer
* No other concurrent cytotoxic investigational drugs
* No concurrent disulfiram

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2005-07; Primary Completion 2005-10 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose
Toxicity
Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Bonny L. Johnson, RN, MSN, Study Chair — Vion Pharmaceuticals
Locations (1):
- M.D. Anderson Cancer Center at University of Texas, Houston, Texas, United States